CLINICAL TRIAL: NCT02722538
Title: A Phase 1b, Multicenter, Open Label Study Evaluating Safety, Tolerability and Preliminary Efficacy of GemRIS 225 mg in Subjects With Muscle-Invasive Transitional Cell Carcinoma of the Bladder
Brief Title: Safety and Tolerability of GemRIS 225 mg in Subjects With Muscle-Invasive Bladder Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taris Biomedical LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAR-200-101
Record Dates: First submitted 2016-02-25; First posted 2016-03-30 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Urinary Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- Residual Tumor following TURBT (Experimental): TAR-200 is placed into the bladder through an inserter on Study Day 0 and is removed on Study Day 7. TAR-200 releases gemcitabine gradually during the 7 day indwelling time. A second TAR-200 is placed in the bladder on Study Day 21 and is removed on Study Day 28, which is the day of the Radical Cystectomy (RC).
  Interventions: Drug: Gemcitabine-Releasing Intravesical System (GemRIS)/TAR-200
- No Residual Tumor Following TURBT (Experimental): TAR-200 is placed into the bladder through an inserter on Study Day 0 and is removed on Study Day 7. TAR-200 releases gemcitabine gradually during the 7 day indwelling time. A second TAR-200 is placed in the bladder on Study Day 21 and is removed on Study Day 28, which is the day of the Radical Cystectomy (RC).
  Interventions: Drug: Gemcitabine-Releasing Intravesical System (GemRIS)/TAR-200

INTERVENTIONS:
Drug: Gemcitabine-Releasing Intravesical System (GemRIS)/TAR-200 — TAR-200 is a passive, nonresorbable gemcitabine-releasing intravesical drug delivery system, regulated as a drug, whose primary mode of action is the controlled release of gemcitabine into the bladder over a 7-day period.

SUMMARY:
The purpose of this study is to determine if TAR-200, an investigational drug-delivery system, is safe and tolerable in patients with muscle-invasive bladder cancer (MIBC) between diagnosis and radical cystectomy (RC).

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of muscle-invasive transitional cell carcinoma of the bladder (stage II-III). Subjects with evidence of metastatic nodal disease to the obuturator or presacral lymph nodes only may be included (N1 M0). Subjects with any degree of fixation of the pelvic sidewall are not eligible.
* In Arm 1, subjects must have residual visible tumor following TURBT. In Arm 2, subjects must be fully resected (i.e., no visible tumor or as little tumor as possible) after restaging TURBT 2-6 weeks prior to Study Day 0.
* Adequate bone marrow, liver, and renal function, as assessed by the following requirements conducted within 21 days prior to dosing:

  1. Hemoglobin ≥ 9.0 g/dL
  2. Absolute neutrophil count (ANC) ≥ 1,500/mm3
  3. Platelet count ≥ 100,000/mm3
  4. Total bilirubin ≤ 1.5xULN (upper limit of normal)
  5. Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 2.5xULN
  6. Glomerular Filtration Rate (GFR) ≥ 30% (≥ 30 ml/min/1.73 m2)
* Subjects must be willing to undergo a cystoscopy on study for investigational product removal.
* Eligible for and willing to undergo RC per the attending urologist.
* Subjects must be deemed ineligible for cisplatin-based combination chemotherapy by the attending medical oncologist.
* Subjects medically eligible for neoadjuvant cisplatin-based combination chemotherapy who refuse this therapeutic option and understand the risks and benefits of doing so.
* Prior radiation therapy is allowed provided that no radiation therapy was administered to the urinary bladder.
* Written informed consent and Health Insurance Portability and Accountability Act of 1966 (HIPAA) authorization for release of personal health information.
* Age > 18 years at the time of consent.

Exclusion Criteria:

* Active malignancies within 12 months with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome.
* Prior systemic chemotherapy for transitional cell carcinoma of the bladder. Any other prior systemic chemotherapy for a non-urothelial carcinoma must have been completed > 5 years prior to initiation of study.
* Previous exposure to gemcitabine instillations.
* Currently receiving other intravesical chemotherapy.
* Concurrent clinically significant infections as determined by the treating investigator.
* Presence of any bladder or urethral anatomic feature that in the opinion of the investigator may prevent the safe placement, indwelling use or removal of TAR-200.
* Documented history of vesicoureteral reflux or the presence of an indwelling ureteral stent or nephrostomy tube at the time of screening.
* Pelvic radiotherapy administered within less than 6 months prior to enrollment. Subjects who received radiotherapy ≥ 6 months prior to enrollment must demonstrate no cystoscopic evidence or symptoms of radiation cystitis.
* Bladder Post-Void Residual Volume (PVR) of > 250-mL.
* Active, uncontrolled urogenital bacterial, viral or fungal infections, including urinary tract infection that in the opinion of the investigator, contraindicates participation. Skin/nail fungal infections are not exclusionary. Subjects with active shingles (varicella zoster infection) will be excluded from the study.
* History or presence of any significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, gynecological, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder that, in the opinion of the investigator, contraindicates participation.
* History of diagnosis of neurogenic bladder.
* Concomitant immunosuppressive medications, such as methotrexate or TNF inhibitors, within 2 weeks of Study Day 0, exclusive of steroid doses ≤ 5 mg daily.
* Difficulty providing blood samples.
* Unwilling or unable to provide informed consent or comply with the requirements of this protocol, including the presence of any condition (physical, mental or social) that is likely to affect the subject's return for scheduled visits and follow-up.
* Other unspecified reasons that, in the opinion of the investigator or TARIS, make the subject unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) coded with MedDRA and graded for severity with CTCAE v4.0 | Maximum 132 days

SECONDARY OUTCOMES:
Number of participants who are tolerant of TAR-200 indwelling | From Day 0 up to Day 7
Percentage of participants who are tolerant of TAR-200 indwelling | From Day 0 up to Day 7
Number of participants who are tolerant of TAR-200 indwelling | From Day 21 up to Day 28
Percentage of participants who are tolerant of TAR-200 indwelling | From Day 21 up to Day 28
Cmax, plasma dFdU | From Day 0 up to Day 28
  Analysis of Cmax (maximum concentration achieved over time) of diflourodeoxyuridine (dFdU) in plasma.
Tmax, plasma dFdU | From Day 0 up to Day 28
  Analysis of Tmax (Day at which maximum concentration was achieved) of diflourodeoxyuridine (dFdU) in plasma.
Cavg, plasma dFdU | From Day 0 up to Day 28
  Analysis of Descriptive statistics (e.g. sample size, mean and median, quartiles, minimum and maximum and box plots) of the concentration of diflourodeoxyuridine (dFdU) in plasma
Cmax, plasma dFdC | From Day 0 up to Day 28
  Analysis of Cmax (maximum concentration achieved over time) of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in plasma
Tmax, plasma dFdC | From Day 0 up to Day 28
  Analysis of Tmax (Day at which maximum concentration was achieved) of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in plasma
Cavg, plasma dFdC | From Day 0 up to Day 28
  Analysis of Descriptive statistics (e.g. sample size, mean and median, quartiles, minimum and maximum and box plots) of the concentration of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in plasma
Cmax, urine dFdU (Arm 1 only) | From Day 0 up to Day 28
  Analysis of Cmax (maximum concentration achieved over time) of diflourodeoxyuridine (dFdU) in urine
Tmax, urine dFdU (Arm 1 only) | From Day 0 up to Day 28
  Analysis of Cmax (maximum concentration achieved over time) of diflourodeoxyuridine (dFdU) in urine
Cavg, urine dFdU (Arm 1 only) | From Day 0 up to Day 28
  Analysis of Descriptive statistics (e.g. sample size, mean and median, quartiles, minimum and maximum and box plots) of the concentration of diflourodeoxyuridine (dFdU) in urine
Cmax, urine dFdC (Arm 1 only) | From Day 0 up to Day 28
  Analysis of Cmax (maximum concentration achieved over time) of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in urine
Tmax, urine dFdC (Arm 1 only) | From Day 0 up to Day 28
  Analysis of Tmax (Day at which maximum concentration was achieved) of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in urine
Cavg, urine dFdC (Arm 1 only) | From Day 0 up to Day 28
  Analysis of Descriptive statistics (e.g. sample size, mean and median, quartiles, minimum and maximum and box plots) of the concentration of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in urine.
Preliminary anti-tumor effects assessed in tumor material (post-treatment) for immunohistochemical tissue biomarkers of drug-induced cell death (AKT) (Arm 1) | Anti-tumor analysis will occur at study visit Day 28.
Preliminary anti-tumor effects assessed in tumor material (post-treatment) for immunohistochemical tissue biomarkers of drug-induced cell death (CD31) (Arm 1) | Anti-tumor analysis will occur at study visit Day 28.
Preliminary anti-tumor effects assessed in tumor material (post-treatment) for immunohistochemical tissue biomarkers of drug-induced cell death (Ki67) (Arm 1) | Anti-tumor analysis will occur at study visit Day 28.
Preliminary anti-tumor effects assessed in tumor material (post-treatment) for immunohistochemical tissue biomarkers of drug-induced cell death (TUNEL) (Arm 1) | Anti-tumor analysis will occur at study visit Day 28.
Preliminary anti-tumor effects assessed in tumor material (post-treatment) for immunohistochemical tissue biomarkers of drug-induced cell death (CD4) (Arm 1) | Anti-tumor analysis will occur at study visit Day 28.
Preliminary anti-tumor effects assessed in tumor material (post-treatment) for immunohistochemical tissue biomarkers of drug-induced cell death (CD8) (Arm 1) | Anti-tumor analysis will occur at study visit Day 28.
Preliminary anti-tumor effects assessed in tumor material (post-treatment) for immunohistochemical tissue biomarkers of drug-induced cell death (PD-L1) (Arm 1) | Anti-tumor analysis will occur at study visit Day 28.
Preliminary anti-tumor effects assessed in tumor material (post-treatment) for immunohistochemical tissue biomarkers of drug-induced cell death (AKT) (Arm 2) | Anti-tumor analysis will occur at study visit Day 42.
Preliminary anti-tumor effects assessed in tumor material (post-treatment) for immunohistochemical tissue biomarkers of drug-induced cell death (CD31) (Arm 2) | Anti-tumor analysis will occur at study visit Day 42.
Preliminary anti-tumor effects assessed in tumor material (post-treatment) for immunohistochemical tissue biomarkers of drug-induced cell death (Ki67) (Arm 2) | Anti-tumor analysis will occur at study visit Day 42.
Preliminary anti-tumor effects assessed in tumor material (post-treatment) for immunohistochemical tissue biomarkers of drug-induced cell death (TUNEL) (Arm 2) | Anti-tumor analysis will occur at study visit Day 42.
Preliminary anti-tumor effects assessed in tumor material (post-treatment) for immunohistochemical tissue biomarkers of drug-induced cell death (CD4) (Arm 2) | Anti-tumor analysis will occur at study visit Day 42.
Preliminary anti-tumor effects assessed in tumor material (post-treatment) for immunohistochemical tissue biomarkers of drug-induced cell death (CD8) (Arm 2) | Anti-tumor analysis will occur at study visit Day 42.
Preliminary anti-tumor effects assessed in tumor material (post-treatment) for immunohistochemical tissue biomarkers of drug-induced cell death (PD-L1) (Arm 2) | Anti-tumor analysis will occur at study visit Day 42.

CONTACTS AND LOCATIONS:
Overall Officials: Siamak Daneshmand, MD, Principal Investigator — University of Southern California
Locations (6):
- United States (5):
  - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Columbia University Medical Center, New York, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
- Radboudumc, Nijmegen, Netherlands

REFERENCES:
- [Derived] Daneshmand S, Brummelhuis ISG, Pohar KS, Steinberg GD, Aron M, Cutie CJ, Keegan KA, Maffeo JC, Reynolds DL, Raybold B, Chau A, Witjes JA. The safety, tolerability, and efficacy of a neoadjuvant gemcitabine intravesical drug delivery system (TAR-200) in muscle-invasive bladder cancer patients: a phase I trial. Urol Oncol. 2022 Jul;40(7):344.e1-344.e9. doi: 10.1016/j.urolonc.2022.02.009. Epub 2022 Apr 14. PMID 35431132